CLINICAL TRIAL: NCT04611490
Title: Comparison of Preoperative 3D Spine Reconstruction With the EOS System and Peroperative 3D Spine Reconstruction With SURGIVISIO
Brief Title: Preoperative and Peroperative Comparison Between 3D Spine Reconstructions
Acronym: Spine-PDCA-OR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.129; 2020-A01071-38 (Other: ID RCB)
Record Dates: First submitted 2020-07-30; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Scoliosis Idiopathic; Navigation, Spatial; Fusion of Spine; Safety Issues
MeSH Terms: conditions — Spatial Navigation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spine Fusion — Each patient will undergo a spine fusion for a evolutive idiopathic scoliosis with the help of the surgivisio system.

SUMMARY:
The objective is to collect data from a per-operative navigation system called SURGIVISIO during scoliosis surgeries. A research program is in progress in order super-impose pre-operative 3D reconstructions of the spine performed with the EOS system on the per-operative 3D reconstructions performed with the SURGIVISIO system.

The purpose of the study is to collect the pre and per operatives data in order to perform the research and development program.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 12 and 20
* Adolescent idiopathic scoliosis
* Fusion surgery planned

Exclusion Criteria:

* Patient under "tutelle" or privation of liberty
* Opposition of parents or patient

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will involve only patients with adolescent idiopathic scoliosis planned for a fusion surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Comparison between the shape of of the spine in supine position in the OR with the Surgivisio system and the 3D shape with the 3D pre-operative planning with the EOS | 1 day
  Comparison in degrees of the pre-operative Cobb angle with the EOS system and the per-operative spine reconstruction with the Surgivisio System.

SECONDARY OUTCOMES:
Vertebrae automatic segmentation in 3D and 2D | 1 year
  The Haussdorff distance will be computed (mm)
Automatic identification of the vertebrae | 1 year
  The Haussdorff distance will be computed (mm)
Evaluation of respiratory movements on image quality | 1 year
  The ratio between respiratory movement and the recalage error (no unit) will be computed
Evaluation of the "recalage" accuracy between preop planning and CBCT perop. | 1 year
  The root mean square error will be computed between the preop and perop 3D shape of the spine.
Evaluation of angular measurements between preop and perop images | 1 year
  Comparison of angular measurements (degrees) of the spine curves between preop and perop images
Evaluation of angular measurements between preop and postop images | 1 year
  Comparison of angular measurements (degrees) of the spine curves between preop and postop images
Evaluation of angular measurements between 1st erect postop Xrays and + 6 months postop Xrays. | 1 year
  Comparison of angular measurements (degrees) of the spine curves between 1s erect postop and 6 months postop images
Evaluation angular measurements between 1st erect postop Xrays and the preop planning | 1 year
  Comparison of angular measurements (degrees) of the spine curves between 1rst erect postop and preop images

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Courvoisier, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubousset J. Scoliosis and its pathophysiology: do we understand it? Spine (Phila Pa 1976). 2001 May 1;26(9):1001. doi: 10.1097/00007632-200105010-00002. No abstract available. PMID 11337615
- [Background] Weinstein SL, Dolan LA, Cheng JC, Danielsson A, Morcuende JA. Adolescent idiopathic scoliosis. Lancet. 2008 May 3;371(9623):1527-37. doi: 10.1016/S0140-6736(08)60658-3. PMID 18456103
- [Background] Courvoisier A, Garin C, Vialle R, Kohler R. The change on vertebral axial rotation after posterior instrumentation of idiopathic scoliosis. Childs Nerv Syst. 2015 Dec;31(12):2325-31. doi: 10.1007/s00381-015-2891-3. Epub 2015 Sep 4. PMID 26337699
- [Background] Merloz P, Tonetti J, Cinquin P, Lavallee S, Troccaz J, Pittet L. [Computer-assisted surgery: automated screw placement in the vertebral pedicle]. Chirurgie. 1998 Nov;123(5):482-90. doi: 10.1016/s0001-4001(99)80077-4. French. PMID 9882919
- [Background] Merloz P, Tonetti J, Pittet L, Coulomb M, Lavallee S, Troccaz J, Cinquin P, Sautot P. Computer-assisted spine surgery. Comput Aided Surg. 1998;3(6):297-305. doi: 10.1002/(SICI)1097-0150(1998)3:63.0.CO;2-8. PMID 10379979
- [Background] Merloz P, Troccaz J, Vouaillat H, Vasile C, Tonetti J, Eid A, Plaweski S. Fluoroscopy-based navigation system in spine surgery. Proc Inst Mech Eng H. 2007 Oct;221(7):813-20. doi: 10.1243/09544119JEIM268. PMID 18019467
- [Background] Prod'homme M, Cavalie G, Kerschbaumer G, Valmary-Degano S, Boudissa M, Tonetti J. T1 Vertebra Pedicular Osteoid Osteoma: Minimally Invasive Surgical Resection Aided by New Integrated Navigation to 3D Imaging Device. Case Rep Orthop. 2019 Mar 18;2019:7626454. doi: 10.1155/2019/7626454. eCollection 2019. PMID 31011459
- [Background] Ferrero E, Mazda K, Simon AL, Ilharreborde B. Preliminary experience with SpineEOS, a new software for 3D planning in AIS surgery. Eur Spine J. 2018 Sep;27(9):2165-2174. doi: 10.1007/s00586-018-5591-3. Epub 2018 Apr 24. PMID 29693200
- [Background] Stindel E, Merloz P, Graf P, Massin P, Gruber P, Robert H, Moineau G, Colmar M. [Computer assisted orthopedics surgery]. Rev Chir Orthop Reparatrice Appar Mot. 2007 Jun;93(4 Suppl):2S11-32. French. PMID 17646826